CLINICAL TRIAL: NCT05660330
Title: Assessing the Effectiveness of a Holistic Semi-tailormade Well-being Intervention at Work: Study Protocol of a Partially Randomized Preference Trial Design
Brief Title: Well-being at Work: Research Into Happiness at Work
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Liantis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: BC10608
Record Dates: First submitted 2022-11-30; First posted 2022-12-21 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Well-being at Work
Keywords: Well-being at work; Work-engagement; Workplace intervention; Holistic; Tailor-made

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holistic semi-tailormade well-being (intervention) group (Experimental): They receive the holistic semi-tailormade intervention, consisting of training and workshops in three well-being domains: psychosocial, ergonomic and lifestyle. In addition to this intervention, they still receive their standard interventions
  Interventions: Behavioral: Holistic semi-tailormade well-being intervention
- Standard well-being (control) group (No Intervention): At first, they receive standard well-being interventions. After six or twelve months, this group can participate in the holistic semi-tailormade well-being intervention.

INTERVENTIONS:
Behavioral: Holistic semi-tailormade well-being intervention — The holistic well-being intervention consists of a mandatory basic package that will take 2 half days and 1 full day to complete. In the first half day, the conclusion of the baseline measurement will be discussed, as well as the specific outline of the well-being thay. On the well-being day, three trained professionals from an HR service company, called Liantis, will guide these interventions (consisting of training and workshops) in the workplace. Only a small proportion of the company employees, called the ambassadors, will attend the well-being day. In the second half day, the ambassadors will be coached to disseminate the obtained information to the entire workplace. This information will be personalized according to the problems, needs and context of each company. Besides the basic package, an optional expertise package will be offered during this second half day. In the period afterwards, the ambassadors are followed every 2 months by means of a semi-structured interview.
  Arms: Holistic semi-tailormade well-being (intervention) group

SUMMARY:
Organizations are becoming increasingly aware that employees are an important factor in gaining and maintaining competitive advantage. Based on the current evidence, a holistic approach, in which different well-being factors and different levels are addressed simultaneously, is needed. However, given the scarcity of this approach in studies, a significant gap in knowledge is demonstrated. This paper tries to address these shortcomings. A partially randomised preference trials design is used to evaluate the impact of an intervention package that focusses on both the individual and organizational level and addresses 3 different domains to improve well-being: psychosocial, ergonomic and lifestyle. The data collection of the research outcomes will be conducted at several points in time. Therefore, a online self-administered questionnaire is developed en will be administered before the start of the intervention. Six and twelve months after the intervention, the short and long term impact of the intervention will be measured. The intervention itself consists of a basic intervention package that will be spread over 3 different days that take place over a time period of maximum 2 weeks. Between 20 and 30 companies will be recruited from a data pool with clients from the Flemish side of Belgium. The sample size of the participating employees should be at least 2000. A stratified random sampling method will be used based on sector type while company size (small-medium-large) will be taken into account

DETAILED DESCRIPTION:
Background

Since there's a high prevalence of people with work-related mental health problems and chronic diseases, the literature used to mainly focus on the negative impact on the well-being of individuals and the consequences for the organizations and how to prevent this.

The last decades, developing methods for preventing health problems has been recognized as crucial and should be high on the agenda of workplace health promotion programs. The introduction of a positive psychology approach to well-being highlights not only the prevention of health problems but especially creating a healthy organization with an environment that can promote employee health and safety as well as organizational effectiveness by enhancing individual and organizational resources .

Organizations are becoming increasingly aware that employees are an important factor in gaining and maintaining competitive advantage . Therefore, literature has seen a growth on research on constructs such as engagement or flow, thriving at work, flourishing at work, meaning at work, and purpose in life or personal growth. Engagement has become one of the most significant concepts in the management field in recent years. It yields positive outcomes such as high levels of well-being and performance . Individuals who are engaged in their work have higher levels of energy, are enthusiastic about their work, and are completely immersed in their work activities. Furthermore, well-being at work is not only crucial for the well-being of the individual employee but it also has positive consequences for the organization, such as better work performance, higher levels of employee creativity and engagement. It has also been associated with lower rates of absenteeism at work.

With most adults spending around half of their waking hours at work, the workplace is an important setting to promote health and well-being. Multiple studies, systematic reviews and meta-analyzes have shown that workplace interventions may result in positive effects. Therefore, it is very important to address and enhance determinants of workplace-related well-being. Interventions that enhance well-being can take place on both the individual level and the organizational level. On the individual level, well-being and health can be improved by different intervention domains. Firstly, physical activity can improve a healthy lifestyle and well-being. Secondly, psychosocial interventions, such as engagement interventions, resilience training or burnout preventions increase mental health and well-being. Lastly, ergonomic interventions, such as sitting behavior has an impact on health . For employees who attended well-being interventions, the number of absence days due to stress, anxiety and depression had fallen over the following three years. In addition, they reported improvements in their relationships, improvements in sleep patterns and improvements in happiness when at work. On the organizational level, workplace well-being programs are expected to reduce employee healthcare costs, increase productivity, and provide a positive return on investment. However, today, empirical evidence for organizational interventions remains limited and the effectiveness of organizational level workplace interventions has not been fully examined. Furthermore, only a small number of studies have thus far examined organizational interventions or activities as potential antecedents of engagement.

It is proven that interventions addressing both the individual and organizational level components simultaneously lead to better results than interventions exclusively focusing on an individual, or an organizational component. Interventions at multiple levels are preferred due to the potential synergistic effects on both employee well-being and performance. Not only is it important to include a combination of both individual-level and organizational-level interventions, but also interventions that are addressing different well-being domains at once - such as ergonomic, psychosocial and lifestyle domain - had a higher chance of reporting significant health improvements than those restricted to one well-being intervention domain. A systematic review indicated that a multi-domain intervention combining physical activity, cognitive training and nutrition exerted beneficial effects. Overall, multi-component programs were more effective than single-component interventions .

Although the monetary aspect (productivity) is an essential part for the organizations whether to implement an intervention or not, organizations and workplaces are also a social and psychological context in which people live, work and relate. Therefore, in order to increase productivity, a holistic intervention approach that addresses more than only the financial aspect, but also other well-being aspects (e.g. engagement and health) will be more effective and should be high on the agenda.

Furthermore, literature has shown the importance of tailor-made interventions because this increases the relevance of the intervention for participants. Tailoring well-being programs have an increased likelihood of success when tailored to the special features of each workplace environment. The effects of the tailored interventions were superior to the generic interventions.

Design

A partially randomized preference trial design with waiting list will be used to assess the effectiveness of an intervention package to improve engagement, job satisfaction and commitment at work. The intervention group will consist of employees from different organizational levels receiving a package of different well-being interventions and will be compared to a control group that does not receive this intervention. Comparison between the groups will be done by collecting psychosocial, ergonomic and lifestyle data through an online questionnaire. The study participants are Flemish adults, employed in a company from one of the following sectors: construction, transportation, industry, IT and health care. We aimed to include at least 2000 participants over 20-30 different companies.

Statistical analysis

Descriptive statistics of baseline characteristics will be reported through numbers and proportions. All analyses will be conducted using SPSS software (version 25.0, SPSS Inc., Chicago, Illinois) or R software (version…., R Core Team…) and the level of significance will be set at p < 0.05 (5%) . T-tests and chi-square tests will be used to compare differences between pre- and post-intervention outcomes and also between intervention participants and non-participants identified at the post-intervention survey.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient knowledge in one of the languages (Dutch, French, English)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Engagement | Change from baseline to post-interventional measurement at 6 and 12 months
  Change in self-reported Utrecht Work Engagement Scale (9 items) from baseline measurement to follow-up measurements at 6 and 12 months
Jobsatisfaction | Change from baseline to post-interventional measurement at 6 and 12 months
  Change in self-reported Jobsatisfaction (1 item) from baseline measurement to follow-up measurements at 6 and 12 months
Commitment | Change from baseline to post-interventional measurement at 6 and 12 months
  Change in self-reported COPSOQ subscale 'Commitment' (5 items) from baseline measurement to follow-up measurements at 6 and 12 months

SECONDARY OUTCOMES:
Life satisfaction | Change from baseline to post-interventional measurement at 6 and 12 months
  Change in self-reported life satisfaction, measured with Cantril Ladder, from baseline measurement to follow-up measurements at 6 and 12 months
Affect | Change from baseline to post-interventional measurement at 6 and 12 months
  Change in self-reported positive and negative affect, measured with the PANAS (10 items), from baseline measurement to follow-ups measurements at 6 and 12 months
Basic needs | Change from baseline to post-interventional measurement at 6 and 12 months
  Change in self-reported basic need satisfaction and frustration, measured with the BNSFS (12 items), from baseline measurement to follow-up measurements at 6 and 12 months
Burnout | Change from baseline to post-interventional measurement at 6 and 12 months
  Change in self-reported burnout, measured with the UBOS (15 items), from baseline measurement to follow-up measurements at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lutgart Braeckman, Principal Investigator — University Ghent; Lieven Annemans, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdin S, Welch RK, Byron-Daniel J, Meyrick J. The effectiveness of physical activity interventions in improving well-being across office-based workplace settings: a systematic review. Public Health. 2018 Jul;160:70-76. doi: 10.1016/j.puhe.2018.03.029. Epub 2018 May 16. PMID 29751224
- [Background] Ahn S, Chung JW, Crane MK, Bassett DR Jr, Anderson JG. The Effects of Multi-Domain Interventions on Cognition: A Systematic Review. West J Nurs Res. 2022 Dec;44(12):1134-1154. doi: 10.1177/01939459211032272. Epub 2021 Jul 14. PMID 34261376
- [Background] Frogeli E, Rudman A, Ljotsson B, Gustavsson P. Preventing stress-related ill health among newly registered nurses by supporting engagement in proactive behaviors: development and feasibility testing of a behavior change intervention. Pilot Feasibility Stud. 2018 Jan 8;4:28. doi: 10.1186/s40814-017-0219-7. eCollection 2018. PMID 29321942
- [Background] Di Fabio A. The Psychology of Sustainability and Sustainable Development for Well-Being in Organizations. Front Psychol. 2017 Sep 19;8:1534. doi: 10.3389/fpsyg.2017.01534. eCollection 2017. PMID 28974935
- [Background] Nielsen, K., Nielsen, M. B., Ogbonnaya, C., Känsälä, M., Saari, E., & Isaksson, K. (2017). Workplace resources to improve both employee well-being and performance: A systematic review and meta-analysis. Work & Stress, 31(2), 101-120.
- [Background] Bakker, A. B., & Albrecht, S. (2018). Work engagement: current trends. Career Development International.
- [Background] Garcia-Buades ME, Peiro JM, Montanez-Juan MI, Kozusznik MW, Ortiz-Bonnin S. Happy-Productive Teams and Work Units: A Systematic Review of the 'Happy-Productive Worker Thesis'. Int J Environ Res Public Health. 2019 Dec 20;17(1):69. doi: 10.3390/ijerph17010069. PMID 31861812
- [Background] Bailey, C., Madden, A., Alfes, K., & Fletcher, L. (2017). The meaning, antecedents and outcomes of employee engagement: A narrative synthesis. International Journal of Management Reviews, 19(1), 31-53.
- [Background] Tandler N, Krauss A, Proyer RT. Authentic Happiness at Work: Self- and Peer-Rated Orientations to Happiness, Work Satisfaction, and Stress Coping. Front Psychol. 2020 Aug 7;11:1931. doi: 10.3389/fpsyg.2020.01931. eCollection 2020. PMID 32849134
- [Background] Kivimaki M, Kawachi I. Work Stress as a Risk Factor for Cardiovascular Disease. Curr Cardiol Rep. 2015 Sep;17(9):630. doi: 10.1007/s11886-015-0630-8. PMID 26238744
- [Background] Vanhove, A. J., Herian, M. N., Perez, A. L., Harms, P. D., & Lester, P. B. (2016). Can resilience be developed at work? A meta-analytic review of resilience-building programme effectiveness. Journal of Occupational and Organizational Psychology, 89(2), 278-307.
- [Background] Awa WL, Plaumann M, Walter U. Burnout prevention: a review of intervention programs. Patient Educ Couns. 2010 Feb;78(2):184-90. doi: 10.1016/j.pec.2009.04.008. Epub 2009 May 20. PMID 19467822
- [Background] Chu AH, Ng SH, Tan CS, Win AM, Koh D, Muller-Riemenschneider F. A systematic review and meta-analysis of workplace intervention strategies to reduce sedentary time in white-collar workers. Obes Rev. 2016 May;17(5):467-81. doi: 10.1111/obr.12388. Epub 2016 Mar 15. PMID 26990220
- [Background] Isham, A., Mair, S., & Jackson, T. (2020). Wellbeing and productivity: a review of the literature.
- [Background] Pieper C, Schroer S, Eilerts AL. Evidence of Workplace Interventions-A Systematic Review of Systematic Reviews. Int J Environ Res Public Health. 2019 Sep 23;16(19):3553. doi: 10.3390/ijerph16193553. PMID 31547516
- [Background] Grant, A. M. (2012). ROI is a poor measure of coaching success: towards a more holistic approach using a well-being and engagement framework. Coaching: An International Journal of Theory, Research and Practice, 5(2), 74-85.
- [Background] Shi Y, Sears LE, Coberley CR, Pope JE. The association between modifiable well-being risks and productivity: a longitudinal study in pooled employer sample. J Occup Environ Med. 2013 Apr;55(4):353-64. doi: 10.1097/JOM.0b013e3182851923. PMID 23567993
- [Background] Noar SM, Benac CN, Harris MS. Does tailoring matter? Meta-analytic review of tailored print health behavior change interventions. Psychol Bull. 2007 Jul;133(4):673-93. doi: 10.1037/0033-2909.133.4.673. PMID 17592961
- [Background] De Cocker K, De Bourdeaudhuij I, Cardon G, Vandelanotte C. The Effectiveness of a Web-Based Computer-Tailored Intervention on Workplace Sitting: A Randomized Controlled Trial. J Med Internet Res. 2016 May 31;18(5):e96. doi: 10.2196/jmir.5266. PMID 27245789
- [Background] Lustria ML, Noar SM, Cortese J, Van Stee SK, Glueckauf RL, Lee J. A meta-analysis of web-delivered tailored health behavior change interventions. J Health Commun. 2013;18(9):1039-69. doi: 10.1080/10810730.2013.768727. Epub 2013 Jun 10. PMID 23750972
- [Background] Brewin CR, Bradley C. Patient preferences and randomised clinical trials. BMJ. 1989 Jul 29;299(6694):313-5. doi: 10.1136/bmj.299.6694.313. No abstract available. PMID 2504416
- [Background] Ivandic I, Freeman A, Birner U, Nowak D, Sabariego C. A systematic review of brief mental health and well-being interventions in organizational settings. Scand J Work Environ Health. 2017 Mar 1;43(2):99-108. doi: 10.5271/sjweh.3616. Epub 2017 Jan 2. PMID 28042963
- [Background] Varekamp I, van Dijk FJ. Workplace problems and solutions for employees with chronic diseases. Occup Med (Lond). 2010 Jun;60(4):287-93. doi: 10.1093/occmed/kqq078. PMID 20511269
- [Background] Woodhouse E, Homewood KM, Beauchamp E, Clements T, McCabe JT, Wilkie D, Milner-Gulland EJ. Guiding principles for evaluating the impacts of conservation interventions on human well-being. Philos Trans R Soc Lond B Biol Sci. 2015 Nov 5;370(1681):20150103. doi: 10.1098/rstb.2015.0103. PMID 26460137
- [Background] Knight C, Patterson M, Dawson J. Building work engagement: A systematic review and meta-analysis investigating the effectiveness of work engagement interventions. J Organ Behav. 2017 Jul;38(6):792-812. doi: 10.1002/job.2167. Epub 2016 Dec 13. PMID 28781428
- [Background] Astrella JA. Return on Investment: Evaluating the Evidence Regarding Financial Outcomes of Workplace Wellness Programs. J Nurs Adm. 2017 Jul/Aug;47(7-8):379-383. doi: 10.1097/NNA.0000000000000499. PMID 28727623
- [Background] Montano D, Hoven H, Siegrist J. Effects of organisational-level interventions at work on employees' health: a systematic review. BMC Public Health. 2014 Feb 8;14:135. doi: 10.1186/1471-2458-14-135. PMID 24507447
- [Background] Knight, C., Patterson, M., & Dawson, J. (2019). Work engagement interventions can be effective: a systematic review. European Journal of Work and Organizational Psychology, 28(3), 348-372.
- [Background] DeChant PF, Acs A, Rhee KB, Boulanger TS, Snowdon JL, Tutty MA, Sinsky CA, Thomas Craig KJ. Effect of Organization-Directed Workplace Interventions on Physician Burnout: A Systematic Review. Mayo Clin Proc Innov Qual Outcomes. 2019 Sep 26;3(4):384-408. doi: 10.1016/j.mayocpiqo.2019.07.006. eCollection 2019 Dec. PMID 31993558
- [Background] Hoek RJA, Havermans BM, Houtman ILD, Brouwers EPM, Heerkens YF, Zijlstra-Vlasveld MC, Anema JR, van der Beek AJ, Boot CRL. Stress Prevention@Work: a study protocol for the evaluation of a multifaceted integral stress prevention strategy to prevent employee stress in a healthcare organization: a cluster controlled trial. BMC Public Health. 2017 Jul 17;18(1):26. doi: 10.1186/s12889-017-4585-0. PMID 28716117
- [Background] Kröll, C., Doebler, P., & Nüesch, S. (2017). Meta-analytic evidence of the effectiveness of stress management at work. European Journal of Work and Organizational Psychology, 26(5), 677-693.
- [Background] Proper KI, van Oostrom SH. The effectiveness of workplace health promotion interventions on physical and mental health outcomes - a systematic review of reviews. Scand J Work Environ Health. 2019 Nov 1;45(6):546-559. doi: 10.5271/sjweh.3833. Epub 2019 May 28. PMID 31134284